CLINICAL TRIAL: NCT06975852
Title: Trauma-Exposed Children and Adolescents: A One-Year Follow-Up Study
Brief Title: Follow-Up Study on Children Exposed to Trauma
Status: Recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Beyza Nur Karal, Research Assistant, MD, Istanbul University
Other Study IDs: 2025/156
Record Dates: First submitted 2025-04-25; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Post-traumatic Stress Disorder (PTSD); Complex Post-Traumatic Stress Disorder (CPTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
As far as it is known, there is no longitudinal study in Turkey investigating the follow-up and treatment of children and adolescents exposed to trauma. This study is planned to reassess children and adolescents with trauma exposure who were evaluated in Istanbul Faculty of Medicine Child Psychiatry outpatient clinic as part of a thesis study one year ago (January-April 2024) and to examine how many of them continue to meet the criteria for Post-Traumatic Stress Disorder (PTSD), how many receive a diagnosis of Complex Post-Traumatic Stress Disorder (CPTSD), and which factors are associated with these outcomes. In this way, it is aimed to contribute to the literature on the long-term effects of trauma exposure. Additionally, since there is no scale in our country that assesses the diagnosis of CPTSD in children, the study also aims to translate the Child and Adolescent Trauma Screen Scale - 2 (CATS-2) into Turkish and examine its psychometric properties.

DETAILED DESCRIPTION:
This study will be conducted under the coordination of Istanbul Faculty of Medicine, Department of Child and Adolescent Psychiatry. Children and adolescents between the ages of 7-18 who have been exposed to trauma and who applied to the Child and Adolescent Psychiatry outpatient clinic of Istanbul Faculty of Medicine and who were evaluated within the scope of the thesis study one year ago (January-April 2024) will be re-evaluated one year later. It is aimed to reach all 210 children and adolescents and evaluate those who agree to participate in the study.

Sample:

* Children-adolescents who were exposed to at least one traumatic event and who were evaluated within the scope of the thesis study one year ago (January-April 2024),
* Children and adolescents aged 7-18,
* Children and/or parents with adequate literacy and Turkish language skills,
* Those without psychotic/manic symptoms or a diagnosis of autism spectrum disorder or intellectual disability in the child or parent during the interview,
* Volunteers who agree to participate in the study.

Researchers will explain the study to volunteer children and their families and present the Informed Consent Form to determine their willingness to participate.

Parents of eligible volunteers will complete the following assessments:

* Sociodemographic Data Form
* Hospital Anxiety and Depression Scale
* Advers Childhood Events Scale
* Positive Childhood Experiences Scale
* Strengths and Difficulties Questionnaire (Parent Form)
* Child and Adolescent Trauma Screen 2 - Caregiver Report

Volunteer children and adolescents will complete:

* Child and Adolescent Trauma Screen 2 - Self Report
* Revised Children's Anxiety and Depression Scale
* Positive Childhood Experiences Scale
* (Adolescent/Child's Self Report) Responses to Stress Questionnaire (Peer Stress)

The clinician will conduct the following assessments:

* ICD-11-based clinical interview
* UCLA PTSD Reaction Index for DSM-5
* Children's Global Assessment Scale (CGAS)

The start date for the study is February 17, 2025, and data analysis will commence afterward. Data will be analyzed using the Statistical Program for Social Sciences (SPSS for Windows, version 21.0). The study is expected to be completed by July 2025.

The coordinating center responsible for the research is the Department of Child and Adolescent Psychiatry at Istanbul Faculty of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Children-adolescents who were exposed to at least one traumatic event and who were evaluated within the scope of the thesis study one year ago (January-April 2024),
* Children and adolescents aged 7-18,
* Children and/or parents with adequate literacy and Turkish language skills.

Exclusion Criteria:

* The presence of psychotic/manic symptoms in the child or parent during the interview or any condition that makes the interview and assessment impossible (e.g., mental or developmental condition or a different communication language),
* The child or parent refusing to participate in the study,
* The presence of autism spectrum disorder or intellectual disability at a severity that prevents assessment.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients applying to the Child and Adolescent Psychiatry outpatient clinic of Istanbul Faculty of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-07-18 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of PTSD and Complex PTSD in Children and Adolescents Exposed to Trauma | Baseline
  This study aims to investigate the prevalence of PTSD and CPTSD diagnoses one year after the initial assessment of trauma-exposed children and adolescents evaluated in our outpatient clinic between January and April 2024 as part of a thesis study.
Factors Associated with the Diagnosis of PTSD and Complex PTSD | Baseline
  We aim to investigate the correlations between PTSD, CPTSD diagnoses and various clinical measures, such as the child's PTSD symptom severity assessed by the UCLA RI-5, the child's PACE score, the parent's ACE and PACE scores, and the severity of parental anxiety and depression.
Adaptation of the Child and Adolescent Trauma Screen - 2 into Turkish, Evaluation of Its Psychometric Properties | Baseline
  Given the absence of an existing instrument to assess CPTSD in children in Turkey, this study also aims to translate the Child and Adolescent Trauma Screen - 2 (CATS-2) into Turkish and to evaluate its psychometric properties. The results of both the self-report and caregiver-report versions of the Turkish CATS-2, completed by children/adolescents and their parents respectively, will be compared with PTSD and CPTSD diagnoses obtained through a clinician-administered ICD-11-based clinical interview, as well as with the results of the UCLA PTSD Reaction Index for DSM-5 (RI-5).

CONTACTS AND LOCATIONS:
Overall Officials: Abdurrahman C Orengul, Associate Professor, Principal Investigator — Istanbul Faculty of Medicine, Child and Adolescent Psychiatry Department
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)